CLINICAL TRIAL: NCT03152578
Title: Randomized, Double Blind, Placebo Controlled Crossover Trial With Open Label Extension Of Topical 20% Beta Caryophyllene Alone And In Combination With 0.025% Capsaicin In The Treatment Of Pain Caused By Osteoarthritis Of The Knee
Brief Title: Topical Use of 20% Beta Caryophyllene Alone And In Combination With 0.025% Capsaicin for Pain Caused by Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Panag Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANAG-001
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BetaC + Capsacian (Active Comparator): 1-3 mls BetaC + Capsacian applied to the painful areas, once upon awakening, once mid day and once before bed-time, each day for two (2) weeks.
  Interventions: Other: BetaC + Capsaicin Topical Cream
- BetaC Only (Active Comparator): 1-3 mls BetaC applied to the painful areas, once upon awakening, once mid day and once before bed-time, each day for two (2) weeks.
  Interventions: Other: BetaC Topical Cream
- Placebo (Placebo Comparator): 1-3 mls Placebo applied to the painful areas, once upon awakening, once mid day and once before bed-time, each day for two (2) weeks.
  Interventions: Other: Placebo Topical Cream

INTERVENTIONS:
Other: BetaC + Capsaicin Topical Cream — BetaC + Capsacin Topical Cream applied to painful knee area 3 times per day.
  Arms: BetaC + Capsacian
Other: BetaC Topical Cream — BetaC Topical Cream Cream applied to painful knee area 3 times per day.
  Arms: BetaC Only
Other: Placebo Topical Cream — Placebo Cream applied to painful knee area 3 times per day.
  Arms: Placebo

SUMMARY:
This study consists of a randomized, double-blind, placebo-controlled crossover trial with open label extension evaluating a topical natural health cream containing ß-caryophyllene alone and in combination with 0.025% capsicum oleoresin against placebo. At the end of the randomized controlled phase of the trial all participants will be given open-label combination cream to be administered over the subsequent 3 weeks.

Primary Endpoint: Evaluation of improvement in pain interference as measured by the BPI in individuals who are experiencing pain due to osteoarthritis of the knee.

Secondary Endpoints: Secondary endpoints are: Confirmation of safety of the topical cream when used daily over 10 weeks.

Further evaluation will include overall patient satisfaction with the products tested.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to American College of Rheumatology criteria: Knee pain with 3 of the following:

  * age >50 years
  * stiffness less than 30 min
  * crepitus,
  * bony tenderness,
  * bony enlargement,
  * no palpable warmth
* Moderate to severe pain, as defined by an average 7-day pain score of greater than 4.0 on an 11-point numerical rating scale for pain intensity (NRS-PI).
* All concurrent medications taken for any reason stable for 14 days
* Ability to follow protocol with reference to cognitive and situational factors (e.g. stable housing, ability to attend visits)
* Ability to read and write English
* Willing and able to give informed consent

Exclusion Criteria:

* Currently using other topical agents for treatment of pain or inflammation
* Use of glucosamine, methysulfonylmethane or other regular anti-inflammatories within 2 weeks prior to completing baseline pain measure and during the trial
* Presence of significant medical disorder that would compromise the participant's safety to take part in the trial (e.g. cancer, immunosuppressed)
* Pregnant and breastfeeding women.
* Type I or Type II diabetes and other endocrine disorders
* Use of exercise or transcutaneous electrical nerve stimulation prior to and during the trial
* A history or present disease (i.e. inflammatory, infectious joint disease) which may affect the outcome of the trial
* Currently taking NHPs for joint health
* Currently enrolled in other clinical trial involving a pharmaceutical treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Score Diary | 2 weeks
  Change in mean daily pain diary score from baseline (average pain score over 7 days pre-treatment) to post treatment

SECONDARY OUTCOMES:
BPI-Short Form | 12 weeks
Patient's Global Impression of Change | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada